CLINICAL TRIAL: NCT00914238
Title: A Randomized Clinical Trial of the Effect of Five-years Versus Two-years Specialized Assertive Intervention for First Episode Psychosis - the OPUS II Trial
Brief Title: Extended Specialized Assertive Intervention for First Episode Psychosis
Acronym: OPUSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other); Region Capital Denmark (Other); Medical Research Council (Other Government); Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Merete Nordentoft, Professor, DMSc., Professor, Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Danish OPUS II trial
Record Dates: First submitted 2009-05-28; First posted 2009-06-04 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: First Episode Psychosis of Schizophrenia and Schizotypal Disorder; Psychotic Disorders; Schizophrenia; Schizoaffective Disorder
Keywords: Randomized clinical trial; first episode psychosis of schizophrenia and schizotypal disorder; rehabilitation; psychosocial; health service research; schizotypal Disorder
MeSH Terms: conditions — Schizotypal Personality Disorder; Psychotic Disorders; Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5 year (Experimental): 5 years OPUS treatment
  Interventions: Behavioral: OPUS 5 years
- 2 years of OPUS treatment (Active Comparator): 2 years OPUS treatment and 3 years of treatment as usual
  Interventions: Behavioral: 2 years OPUS treatment

INTERVENTIONS:
Behavioral: 2 years OPUS treatment — 2 years OPUS and transfer to standard treatment.
  Arms: 2 years of OPUS treatment
Behavioral: OPUS 5 years
  Arms: 5 year

SUMMARY:
In a randomized clinical trial, the researchers want to investigate if the positive short-term outcomes (first 1-2 years), achieved with specialized assertive intervention programme (OPUS), can be maintained for five years if the specialized treatment is sustained over the first five years in comparison to only two years of specialized treatment followed by three years of standard treatment.

DETAILED DESCRIPTION:
The Danish OPUS I trial succeeded in randomizing 547 patients with first-episode psychosis to a two-year specialized intensive treatment program (OPUS) or standard treatment. The results clearly favored OPUS treatment, and psychotic and negative symptoms, substance abuse, adherence to treatment, use of anti-psychotic medication, user satisfaction, and use of bed days were better in OPUS compared to standard treatment. However, the five-year follow-up, three years after patients from OPUS were transferred to standard treatment, showed that the positive clinical effects were not sustained, when the intensive treatment was terminated, except from OPUS-patients being less likely to stay in institutions than patients who received standard care.

Objective: The aim in OPUS II trial is to compare the effect of five-years versus two-years specialized assertive intervention program (OPUS-treatment) for first episode psychosis on clinical symptoms, substance abuse, institutionalization, and labor market affiliation.

Hypothesis: It is possible to maintain the positive results of the intensive two-year intervention in another three years for those who keep receiving the specialized assertive intervention program.

Design: Open label randomized clinical trial. Setting: Psychiatric Center Bispebjerg and Center for Psychiatric Research Aarhus, Denmark.Participants: 400 patients with first episode of schizophrenia spectrum disorder received treatment in one of the six OPUS - teams for 1½ years.

Intervention: Another 3½ years OPUS-treatment versus ½ year OPUS-treatment and thereafter referral to standard treatment. The extended OPUS treatment consist modified assertive case management, rational pharmacotherapy, family psycho-educational intervention, group interventions to aid with recovery, social skills training, cognitive behavior therapy when indicated, and crisis intervention. OPUS-treatment is tailored to meet the individual patient's needs.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 - 37 years
* first episode psychosis in schizophrenia spectrum
* treated for 1½ year in the five OPUS teams in the Capital Region and the OPUS teams in Region Midt
* patients who will give signed informed consent to participate in the trial

Exclusion Criteria:

* patients who are not treated in one of the OPUS team in the Capital Region and Region Midt
* patients who don't give signed informed consent to participate in the study

Ages: 18 Years to 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2009-07; Primary Completion 2015-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Negative symptoms, measured with Schedule for Assessment of Negative Symptoms in Schizophrenia, (SANS) | 3 years

SECONDARY OUTCOMES:
Psychotic symptoms | 3 years
Simultaneous remission of both psychotic and negative symptoms. | 3 years
Substance abuse. | 3 years
Suicidal behaviour. | 3 years
Use of bed days. | 3 years
Independent living. | 3 Years
Labour market affiliation. | 3 years
User satisfaction. | 3 years
Adherence to treatment. | 3 years
Compliance with medication | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, Professor, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Psychiatric Center Bispebjerg, Copenhagen
  - Psychiatric Centre Bispebjerg, Copenhagen

REFERENCES:
- [Derived] Puntis S, Minichino A, De Crescenzo F, Cipriani A, Lennox B, Harrison R. Specialised early intervention teams (extended time) for recent-onset psychosis. Cochrane Database Syst Rev. 2020 Nov 2;11(11):CD013287. doi: 10.1002/14651858.CD013287.pub2. PMID 33135812
- [Derived] Albert N, Randers L, Allott K, Jensen HD, Melau M, Hjorthoj C, Nordentoft M. Cognitive functioning following discontinuation of antipsychotic medication. A naturalistic sub-group analysis from the OPUS II trial. Psychol Med. 2019 May;49(7):1138-1147. doi: 10.1017/S0033291718001836. Epub 2018 Jul 30. PMID 30058511
- [Derived] Albert N, Melau M, Jensen H, Emborg C, Jepsen JR, Fagerlund B, Gluud C, Mors O, Hjorthoj C, Nordentoft M. Five years of specialised early intervention versus two years of specialised early intervention followed by three years of standard treatment for patients with a first episode psychosis: randomised, superiority, parallel group trial in Denmark (OPUS II). BMJ. 2017 Jan 12;356:i6681. doi: 10.1136/bmj.i6681. PMID 28082379
- [Derived] Melau M, Harder S, Jeppesen P, Hjorthoj C, Jepsen JR, Thorup A, Nordentoft M. The association between working alliance and clinical and functional outcome in a cohort of 400 patients with first-episode psychosis: a cross-sectional study. J Clin Psychiatry. 2015 Jan;76(1):e83-90. doi: 10.4088/JCP.13m08814. PMID 25650684
- [Derived] Melau M, Jeppesen P, Thorup A, Bertelsen M, Petersen L, Gluud C, Krarup G, Nordentoft M. The effect of five years versus two years of specialised assertive intervention for first episode psychosis - OPUS II: study protocol for a randomized controlled trial. Trials. 2011 Mar 10;12:72. doi: 10.1186/1745-6215-12-72. PMID 21392377